CLINICAL TRIAL: NCT05851183
Title: A Prospective, Open-label, Pragmatic Randomized Controlled Trial to Demonstrate the Effect of Improving the Venous Reflux Time by Vitis Vinifera Seed Extract in Patients With Varicose Vein of Lower Extremity
Brief Title: Effect of Vitis Vinifera Seed Extract on Venous Reflux Time in Varicose Vein
Acronym: VICTORY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, In Hyun Jung, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICTORY trial
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Varicose Veins of Lower Limb

STUDY DESIGN:
Intervention Model Description: The investigators aim to compare and evaluate the improvement effects on venous reflux time in patients with lower extremity varicose veins between lifestyle modifications and the combined treatment of Vitis Vinifera seed extract (Entelon®) administration and lifestyle modifications.
Masking Description: The study is designed as an open-label trial to investigate the efficacy of vitis vinifera extract compared to a group undergoing lifestyle modification alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic lifestyle change (Active Comparator): Therapeutic lifestyle change only
  Interventions: Behavioral: Therapeutic lifestyle change only
- Therapeutic lifestyle change plus Vitis Vinifera extract therapy (Experimental): Therapeutic lifestyle change plus Vitis Vinifera extract medication therapy
  Interventions: Drug: Vitis Vinifera seed extract medication plus therapeutic lifestyle change

INTERVENTIONS:
Drug: Vitis Vinifera seed extract medication plus therapeutic lifestyle change — Administer 150mg of Vitis Vinifera seed extract (Entelon®) orally twice a day
  Other Names: Entelon® medication plus therapeutic lifestyle change
  Arms: Therapeutic lifestyle change plus Vitis Vinifera extract therapy
Behavioral: Therapeutic lifestyle change only — Implementing TLCs is a critical component of a comprehensive treatment plan for varicose veins. A key aspect of TLCs is the optimization of postural habits. Patients are advised to avoid extended sitting or standing periods, which exert additional pressure on the venous system in the lower extremities and exacerbate venous insufficiency. During rest periods, elevating the legs closer to the heart is recommended because this simple yet effective adjustment promotes venous return and reduces the gravitational burden on the venous valves of the legs. The use of graduated compression stockings during waking hours is another therapeutic lifestyle intervention that is often prescribed for patients with varicose veins. Additional TLCs include maintaining optimal body weight and engaging in regular physical exercise Walking or cycling are often recommended because of their effectiveness in promoting lower limb venous return.
  Arms: Therapeutic lifestyle change

SUMMARY:
The number of patients with lower extremity varicose veins has been increasing due to an aging population, with treatments divided into conservative and invasive methods. Current treatments can be expensive and inaccessible for some patients. Entelon, a relatively inexpensive intravenous drug, has shown promise in improving symptoms related to venous lymphatic dysfunction, but its objective vascular function improvement hasn't been proven. This study aims to assess the effectiveness of Vitis Vinifera seed extract (Entelon®) combined with lifestyle therapy in patients with varicose veins, using follow-up Doppler ultrasonography to measure venous reflux improvement.

DETAILED DESCRIPTION:
Varicose veins in the lower extremities are more than the function of the valve membranes on the inside of the legs, and the heart cannot function, resulting in regurgitation in the lower half of the body. This causes blood to pool in the lower extremities and causes various symptoms. Large stalks of superficial veins and venous valves of deep veins become dysfunctional, resulting in an increase in blood vessels in the calf area with backflow of blood. The valvular insufficiency of lower extremity veins is the main cause. In general, it occurs in the great saphenous vein that flows into the deep vein from the groin, the small saphenous vein in the posterior leg, and the perforating vein in the calf. Reflux in superficial veins (e.g. great saphenous vein, small saphenous vein) and deep veins can generally be confirmed using Doppler ultrasound. Determine the direction of treatment by confirming if there is branch vein dilatation. Ultrasonography is also done on the opposite, unaffected side, even if symptoms are in only one leg.

Treatment of varicose veins can generally be divided into conservative treatment and invasive treatment, and lifestyle correction and wearing compression stockings are recommended as conservative treatment. Surgical treatment is indicated when conservative treatment is ineffective or interferes with daily life. Symptoms can be alleviated by removing superficial veins with regurgitation due to valvular insufficiency, or by inducing hardening of the causative blood vessels using high frequency or laser to block regurgitation and prevent blood flow.

However, most of these treatments are non-salary items, and are relatively expensive treatment methods that impose a large financial burden on patients. In addition, deep veins are responsible for 90% of blood transport, but surgical treatment is impossible and only conservative treatment is possible.

As a non-invasive treatment, which is an intravenous active agent, is registered as a drug to be administered, and improvement of symptoms related to venous lymphatic dysfunction (pain, lower extremity anxiety symptoms) is attracting attention. It is relatively inexpensive compared to surgical treatment, but until now, objective improvement of vascular function by drug treatment has not been proven. Vitis Vinifera seed extract (Entelon®) was launched in 1998 and its safety has already been confirmed, and the investigators have investigated the effect of lower limit volume reduction compared to placebo after administration of Vitis Vinifera seed extract in patients with edema. (Sano A, Tokutake S, Seo A. Proanthocyanidin-rich grape seed extract reduces leg swelling in healthy women during prolonged sitting. J Sci Food Agric. 2013 Feb;93(3):457-62.).

In this study, along with lifestyle therapy in patients with varicose veins, follow-up Doppler ultrasonography after administration of Entelon will be used to confirm the improvement effect of venous reflux.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aged between 19 and under 80 years old
2. Patients with the following findings on venous Doppler ultrasound examination:

   * Superficial veins (such as the great saphenous vein, small saphenous vein, etc.) showing valvular reflux for 0.5 seconds or longer
   * Deep veins (such as the femoral vein, etc.) showing valvular reflux for 1 second or longer
3. Patients who have completed the washout period as described below by Visit 2, including the screening period:

   * Analgesics, steroids, anti-inflammatory drugs, and venoactive medications (such as Entelon, etc.): at least 4 weeks
4. Patients who voluntarily provide written informed consent to participate in this clinical trial

Exclusion Criteria:

1. Peripheral arterial occlusive disease in the lower limbs
2. Asymptomatic lower extremity varicose veins
3. Acute deep vein thrombosis
4. Frequent lower limb pain due to neuropathy
5. Patients who have undergone or are scheduled for varicose vein procedures/surgeries (However, patients who have had a procedure or surgery more than 1 year prior to the screening date are eligible to participate)
6. Patients diagnosed with systemic diseases causing edema or thrombosis, such as heart failure, endocrine diseases (hypothyroidism, Cushing's syndrome, uncontrolled diabetes), allergic reactions to medications, urticaria and angioedema, malabsorption and protein-calorie malnutrition, obstructive sleep apnea, or thrombophilia, as determined by the investigator
7. History of malignancy within the past 5 years, but the following cases are eligible for clinical trial participation:

   * Those who have a history within the past 5 years but maintain a cured state without recurrence or metastasis
   * Those who have completed treatment for their tumor and have been disease-free for at least 5 years from the screening date
   * Those who have passed at least 1 year since the screening date after complete resection of basal cell carcinoma/squamous cell carcinoma, radical resection of thyroid papillary cancer, or successful treatment of cervical intraepithelial neoplasia
8. Severe renal dysfunction (serum creatinine levels more than twice the normal upper limit of the institution) at the screening date
9. Severe liver dysfunction (ALT or AST levels more than three times the normal upper limit of the institution) at the screening date
10. Need to receive diuretics or contraindicated medications and therapies that may affect the results of this clinical trial during the study period (However, patients who have been taking antihypertensive medications (calcium channel blockers, beta-blockers, angiotensin-converting enzyme inhibitors, vasodilators, vasoconstrictors) at the same dosage for at least 4 weeks (28 days) before screening and will maintain the same dosage and administration during the study period are eligible to participate)
11. History of clinically significant psychiatric disorders or alcohol abuse
12. History of hypersensitivity reactions to the investigational drug or its ingredients
13. Those who have participated in or are scheduled to participate in other clinical trials (investigational drugs, medical devices, health functional foods) within 12 weeks from the screening date
14. Pregnant or breastfeeding women
15. Women of childbearing potential who plan to become pregnant during the clinical trial participation period
16. Individuals deemed unsuitable for participation in the clinical trial by the investigator

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in venous reflux time | 6, 12 weeks
  The investigators will assess the changes in venous reflux time using lower limb venous Doppler ultrasound examinations. The examination will be performed by an independent assessor who is not aware of the group assignments to ensure unbiased assessment and measurement.

SECONDARY OUTCOMES:
Improvement of venous reflux | 6, 12 weeks
  The investigators will assess the improvement of venous reflux of target vessel (superficial vein < 0.5 seconds, deep vein < 1 seconds)
Change in varicose vein size area | 6, 12 weeks
  The investigators will assess changes in varicose vein diameters using lower-limb venous Doppler ultrasound examinations
Change in venous reflux volume | 6, 12 weeks
  The investigators will assess the changes in venous reflux volume using Venous Doppler Reflux VTI × varicose vein size area
Change of extracellular water ratio | 6, 12 weeks
  The investigators will assess the changes in extracellular water (ECW) ratio (ECW/total body water) of target limb using body composition analyzer (ACCUNIQ BC720®).
Improvement in Venous Clinical Severity Score (VCSS) | 6, 12 weeks
  The Venous Clinical Severity Score (VCSS) assesses the severity of chronic venous diseases. The score ranges from 0 (no symptoms) to 30 (severe venous disease). The scoring system considers various factors, including pain; varicose veins; venous edema; skin pigmentation; inflammation; induration; and active ulcers and their duration, size, and number. A higher VCSS indicates a worse outcome, implying a more severe state of venous disease.
Improvement of 14-item Chronic Venous Insufficiency quality of life Questionnaire (CIVIQ-14) | 6, 12 weeks
  The Chronic Venous Insufficiency Quality of Life Questionnaire (CIVIQ-14) is a valuable tool designed to evaluate the impact of chronic venous insufficiency on quality of life. Improvement in the CIVIQ-14 refers to the enhancement in scores, indicating better management of symptoms, greater comfort, and overall well-being of the patient over the course of treatment or intervention.

CONTACTS AND LOCATIONS:
Overall Officials: In Hyun Jung, MD, PhD, Principal Investigator — Yongin Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yongin Severance Hospitall, Yonsei University College of Medicine, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Gloviczki P, Lawrence PF, Wasan SM, Meissner MH, Almeida J, Brown KR, Bush RL, Di Iorio M, Fish J, Fukaya E, Gloviczki ML, Hingorani A, Jayaraj A, Kolluri R, Murad MH, Obi AT, Ozsvath KJ, Singh MJ, Vayuvegula S, Welch HJ. The 2022 Society for Vascular Surgery, American Venous Forum, and American Vein and Lymphatic Society clinical practice guidelines for the management of varicose veins of the lower extremities. Part I. Duplex Scanning and Treatment of Superficial Truncal Reflux: Endorsed by the Society for Vascular Medicine and the International Union of Phlebology. J Vasc Surg Venous Lymphat Disord. 2023 Mar;11(2):231-261.e6. doi: 10.1016/j.jvsv.2022.09.004. Epub 2022 Oct 12. PMID 36326210
- [Background] Labropoulos N, Tiongson J, Pryor L, Tassiopoulos AK, Kang SS, Ashraf Mansour M, Baker WH. Definition of venous reflux in lower-extremity veins. J Vasc Surg. 2003 Oct;38(4):793-8. doi: 10.1016/s0741-5214(03)00424-5. PMID 14560232
- [Background] Labropoulos N, Leon LR Jr. Duplex evaluation of venous insufficiency. Semin Vasc Surg. 2005 Mar;18(1):5-9. doi: 10.1053/j.semvascsurg.2004.12.002. PMID 15791546
- [Background] De Maeseneer MG, Kakkos SK, Aherne T, Baekgaard N, Black S, Blomgren L, Giannoukas A, Gohel M, de Graaf R, Hamel-Desnos C, Jawien A, Jaworucka-Kaczorowska A, Lattimer CR, Mosti G, Noppeney T, van Rijn MJ, Stansby G, Esvs Guidelines Committee, Kolh P, Bastos Goncalves F, Chakfe N, Coscas R, de Borst GJ, Dias NV, Hinchliffe RJ, Koncar IB, Lindholt JS, Trimarchi S, Tulamo R, Twine CP, Vermassen F, Wanhainen A, Document Reviewers, Bjorck M, Labropoulos N, Lurie F, Mansilha A, Nyamekye IK, Ramirez Ortega M, Ulloa JH, Urbanek T, van Rij AM, Vuylsteke ME. Editor's Choice - European Society for Vascular Surgery (ESVS) 2022 Clinical Practice Guidelines on the Management of Chronic Venous Disease of the Lower Limbs. Eur J Vasc Endovasc Surg. 2022 Feb;63(2):184-267. doi: 10.1016/j.ejvs.2021.12.024. Epub 2022 Jan 11. No abstract available. PMID 35027279
- [Background] AIUM Practice Parameter for the Performance of a Peripheral Venous Ultrasound Examination. J Ultrasound Med. 2020 May;39(5):E49-E56. doi: 10.1002/jum.15263. Epub 2020 Mar 12. No abstract available. PMID 32162338

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT05851183/Prot_SAP_ICF_001.pdf